CLINICAL TRIAL: NCT00169169
Title: Randomised Phase 3 Study of Rituximab in High-Risk Patients With Diffuse Large B-Cell Lymphoma Who Received a First-Line Consolidative Chemotherapy With Autologous Stem Cell Transplant (ASCT).
Brief Title: Efficacy Study of Rituximab After ASCT in High-Risk Diffuse Large B-Cell Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNH-98.3
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: CD20-Positive Large B-Cell Lymphoma
Keywords: Diffuse large B cell lymphoma; Rituximab; Autotransplant
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

INTERVENTIONS:
Drug: ACVBP
Drug: ACE
Drug: rituximab
Procedure: Autologous stem cell transplant

SUMMARY:
Rituximab vs observation after high-dose consolidative first-line chemotherapy (HDC) with autologous stem cell transplantation in poor risk diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This is a multicentric, open-label, randomized clinical study, evaluating the efficacy and the safety of Rituximab After ASCT in patients aged 18 to 59 years with previously untreated High-Risk (aa-IPI 2 or 3 ) Diffuse Large B-Cell Lymphoma .

The duration of the treatment period is approximately 25 weeks and patients are followed until Death.

From 10/99 to 05/03, 476 patients were enrolled. 235 patients were assigned to receive ACE and 241 to ACVBP. Among the 331 patients, in Complete response (CR+CRu) after induction, who received HDC, 269 were randomized (R2) after hematological recovery to receive either rituximab (n=139) or nothing (n=130).

The final analysis was performed in June 2005.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B cell lymphoma (WHO Classification).
* Aged from 18 to 59 years, eligible for transplant.
* Patient not previously treated.
* Age adjusted International Prognostic Index equal to 2 or 3.
* Having previously signed a written informed consent.
* Women of childbearing potential currently practicing an adequate method of contraception.

Exclusion Criteria:

* Any other histological type of lymphoma.
* Any history of treated or non-treated indolent lymphoma.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug contained in the chemotherapy regimens.
* Poor renal function (creatinin level>150mmol/l), poor hepatic function (total bilirubin level>30mmol/l, transaminases>2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils < 1.5 G/l or platelets < 100 G/l, unless related to bone marrow infiltration.
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Any serious active disease (according to the investigator's decision).
* HIV, HTLV1 or HBV related disease.
* Any organ transplantation before inclusion.
* Pregnant women.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 430
Dates: Start 1999-10; Study Completion 2005-08

PRIMARY OUTCOMES:
- To compare event-free survival of patients randomized to receive Rituximab or no further therapy after HDT

SECONDARY OUTCOMES:
- To compare response rate to induction treatments (ACVBP vs AC/ACE).
- To evaluate response rate at the end of treatment.
- To compare overall survival (ACVBP vs AC/ACE; Rituximab / nothing)
- To evaluate the safety and tolerability of Rituximab

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Haioun, Study Chair — Hôpital Henri Mondor, Créteil, France
Locations (5):
- France (5):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - CHRU de Nancy Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Haioun C, Lepage E, Gisselbrecht C, Salles G, Coiffier B, Brice P, Bosly A, Morel P, Nouvel C, Tilly H, Lederlin P, Sebban C, Briere J, Gaulard P, Reyes F. Survival benefit of high-dose therapy in poor-risk aggressive non-Hodgkin's lymphoma: final analysis of the prospective LNH87-2 protocol--a groupe d'Etude des lymphomes de l'Adulte study. J Clin Oncol. 2000 Aug;18(16):3025-30. doi: 10.1200/JCO.2000.18.16.3025. PMID 10944137
- [Background] Coiffier B, Haioun C, Ketterer N, Engert A, Tilly H, Ma D, Johnson P, Lister A, Feuring-Buske M, Radford JA, Capdeville R, Diehl V, Reyes F. Rituximab (anti-CD20 monoclonal antibody) for the treatment of patients with relapsing or refractory aggressive lymphoma: a multicenter phase II study. Blood. 1998 Sep 15;92(6):1927-32. PMID 9731049
- See also: Official site of the Groupe d'Etude des Lymphomes de l'Adulte (In french) — http://www.gela.org